CLINICAL TRIAL: NCT06961825
Title: The Role of Nutrition in the Rehabilitation of Patients With Eating Disorders After a Vascular Stroke: A Randomized Controlled Trial Investigating the Effect of Protein Supplementation on Functional Recovery, Sarcopenia, Osteopenia, and Nutritional Status in Stroke Patients With Hypoalbuminemia.
Brief Title: Brief Title: The Role of Nutrition in the Rehabilitation of Patients With Eating Disorders After a Vascular Stroke.
Acronym: Nutristroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistan Professor of PMR,Orthopaedic Spine Surgeon, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Ioannina
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Hypoalbuminemia; Sarcopenia; Osteopenia; Malnutrition (Calorie); Protein-energy Malnutrition; Functional Decline
Keywords: protein supplementation; nutritional intervention; albumin levels; stroke; stroke rehabilitation; eating disorders; malnutrition; nutritional assessment; sarcopenia; osteopenia
MeSH Terms: conditions — Stroke; Hypoalbuminemia; Sarcopenia; Bone Diseases, Metabolic; Malnutrition; Protein-Energy Malnutrition; Feeding and Eating Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protein Supplement - Single Dose (Experimental): Participants in this arm will receive one dose of protein supplement daily.
  Interventions: Dietary Supplement: Dietary Supplement
- Protein Supplement - Double Dose (Experimental): Participants in this arm will receive two doses of protein supplement daily.
  Interventions: Dietary Supplement: Dietary Supplement
- Control group (No Intervention): no protein supplementation

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — complete, semi-elemental formula for tube feeding and orla intake based on peptides, in powder form, low in fat (32% of energy), high in MCTs (>90% of total fat) free of fiber and gluten
  Arms: Protein Supplement - Double Dose; Protein Supplement - Single Dose

SUMMARY:
Brief Summary: The main objective of this thesis is to investigate the role of nutrition - specifically the administration of protein supplements (single dose and double dose) - in the rehabilitation of stroke patients with low albumin levels in relation to sarcopenia, osteopenia and functional recovery indices. The study will follow a randomized controlled trial design, incorporating clinical observation, analysis of biochemical markers, and assessment of physical and functional parameters. Participants will be randomly assigned to one of the three groups: (1) Group 1, receiving no protein supplementation (control group), (2) Group 2, receiving a single dose of protein supplement and (3) Group 3, receiving a double dose of protein supplement. The intervention will last for at least six weeks or until the biochemical markers of albumin normalize and the patient resumes regular oral intake. Biochemical assessment with be conducted through regular nutritional evaluations including measurement of serum albumin, prealbumin, C - reactive protein, creatinine, blood glucose and glycosylated hemoglobin (HbA1c), urea, electrolytes, urine albumin and additional inflammatory markers. Bone density will be assessed using DEXA, MBSR and hip measurements to determine the potential improvements resulting from the intervention. Muscle mass will be evaluated using whole - body DEXA analysis, while muscle strength and mobility will be assessed through grip strength tests and fine gait assessments. Functional recovery will be evaluated usings standardized tools for activities of daily living (Barthel Index), mental state (Geriatric Depression Scale) and quality of life (SF - 36), as well as mobility and walking tests such as the Timed Up and Go Test and 6 - Minute Walk Test. The collected data will be analyzed using appropriate statistical tools, including comparison models (ANOVA, Mann - Whitney U test) and correlation models (Pearson - Spearman). This research is expected to enhance theoretical knowledge regarding the relationship between nutrition, biochemical markers and rehabilitation outcomes in stroke patients with hypoalbuminemia. More specifically, it aims to explore the underlying mechanisms through which nutrition affects recovery - a field that remains unexplored. Additionally, the anticipated finding may contribute to the development of clinical guidelines and therapeutic approaches for the nutritional management of patients with low albumin levels, promoting personalized nutritional strategies that support effective post - stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Adults aged 18 to 85 years
* Diagnosis: Patients diagnosed with a stroke (cerebrovascular accident) within the last 4 to 6 weeks
* Serum albumin levels: Patients with low serum albumin levels (< 3.5 g / dL)
* Nutritional intervention requirement: Patients who require nutritional intervention to support rehabilitation and nutrition
* Informed consent: Patients who have completed the consent form for participation in the study and acceptance of the intervention

Exclusion Criteria:

* Severe infections or serious cardiopulmonary conditions: Patients with severe infections or serious cardiopulmonary conditions requiring immediate medical intervention, which may affect nutrition and rehabilitation
* Comorbidities: Patients with comorbid conditions such as renal or liver disease
* History of stroke or neurological conditions: Patients with a history of stroke or other neurological conditions who do not meet the criteria for rehabilitation
* Severe mental or psychological conditions: Patients with severe mental or psychological conditions who are unable to understand or consent to participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2030-05-05 (Estimated); Study Completion 2030-05-05 (Estimated)

PRIMARY OUTCOMES:
Serum Albumin Levels | Baseline and every 2 weeks for up to 6 weeks
  Change in serum albumin concentration to assess nutritional status and response to protein supplementation.

SECONDARY OUTCOMES:
Muscle Mass (Whole-body DEXA) | Baseline and at week 6
  Evaluation of changes in muscle mass using DEXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Avraam Ploumis, Principal Investigator — University Hospital, Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece, Greece

IPD SHARING:
Plan to Share IPD: No